CLINICAL TRIAL: NCT01831856
Title: Efficacy and Safety Study of F373280 for Maintenance of Sinus Rhythm After Electrical Cardioversion in Patients With Persistent Atrial Fibrillation and Chronic Heart Failure. International, Multicentric, Randomised, Double-blind, Placebo Controlled Study.
Brief Title: Efficacy and Safety Study of F373280
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F373280 CA 2 01; 2012-003487-48 (EudraCT Number)
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Atrial Fibrillation
Keywords: Cardiovascular diseases; Chronic Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- F373280 (Experimental)
  Interventions: Drug: 1g of F373280
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 1g of F373280 — Oral administration, one capsule each evening with dinner.
  Arms: F373280
Drug: Placebo — Oral administration, one capsule each evening with dinner.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of F373280 on the maintenance of normal cardiac rhythm after direct electric cardioversion in patients with persistent atrial fibrillation and cardiac failure.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged more than 18 years (inclusive)
* Patients with current episode of persistent Atrial Fibrillation (AF) between 7 days and 6 months duration for whom electrical cardioversion is warranted
* Previous history of first documented episode of persistent AF.
* Previous history of ischemic or non ischemic heart failure
* New York Heart Association (NYHA) class I or II chronic heart failure at selection and at inclusion
* Left ventricular systolic dysfunction defined at selection and at inclusion by a reduced left ventricular ejection fraction (LVEF) ≥ 30% and ≤ 45% or for patients with a LVEF > 45%:

  * an increased left ventricular end-diastolic size (diameter ≥ 60 mm and/or > 32 mm/m² and/or volume > 97 ml/m²)
  * and/or an increased left ventricular end-systolic size (diameter > 45 mm and/or > 25 mm/m² and/or volume > 43 ml/m²)
  * and/or a reduced left ventricular outflow tract velocity time integral < 15 cm
* On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers
* Left atrial area ≤ 40 cm² at selection and at inclusion
* Patients treated or having to be treated by vitamin K antagonist
* For female patient of child-bearing potential:

  * In all the countries except Italy:
* Use of an effective method of contraception (hormonal contraception or intra-uterine device) assessed by the investigator, for at least 2 months before the selection in the study, and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment
* Documented as surgically sterilized

  * In Italy only:
* Absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or
* Use of double barrier contraception method (use of effective medical contraception method) from at least 2 months before the start of the study to the entire duration of the study and for a month after the end of the study or
* Documented as surgically sterilized.
* For female patient of child-bearing potential: negative urine pregnancy test at inclusion
* For male with a child-bearing potential partner (In Italy only):
* Absolute abstention from sexual intercourse during the whole duration of the study and for 3 months after the end of the study or
* Use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to 3 months after the end of the study.

Ethical / legal considerations:

* Having signed his/her written informed consent,
* Affiliated to a social security system, or is beneficiary (if applicable in the national regulation)

Exclusion Criteria:

* No previous history of first documented episode of persistent AF
* More than two successful cardioversions (electrical or pharmacological) in the last 6 months
* Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV)
* NYHA class III or IV heart failure at selection or at inclusion
* Thyroid disease uncontrolled by treatment: TSH ± T4L ± T3L to be checked in case of treatment for thyroid disease
* Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection
* Severe chronic kidney disease (creatinine ≥ 25 mg/L or estimated glomerular filtration rate < 30 ml/min) at selection
* Bradycardia (HR ≤ 50 bpm)
* Hyperkalemia or hypokalemia (according to the standards of local laboratories) at selection
* Cardiac surgery within 3 months before selection or planned during the study duration

Criteria related to treatments:

* Previously ineffective pharmacological or electrical cardioversion
* Concomitant treatment with ranolazine or any antiarrhythmic drug (within 7 days prior to selection), except amiodarone, dronedarone and stable dose of digoxin, betablockers, calcium-blockers
* Concomitant treatment with oral amiodarone or dronedarone from selection
* Concomitant treatment with intravenous amiodarone from selection
* Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months
* Treatment with any Polyunsaturated Fatty Acid (PUFA) within the last 3 months
* Dietary supplement with ω 3 or ω 6 according to investigator's judgement
* Having undergone any form of ablation therapy for AF
* Patient treated with oral anticoagulant treatment other than vitamin K antagonist: new oral anticoagulants (dabigatran, rivaroxaban, apixaban), or treated with irreversible antiplatelet agents P2Y12 inhibitors such as ticlopidine, clopidogrel or prasugrel

Other criteria:

* Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion
* Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection
* Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself/herself to its constraints
* Patient family member or work associate (secretary, nurse, technician,..) of the Investigator
* Patient having forfeited his / her freedom by administrative or legal award or being under guardianship
* Breastfeeding female patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karim Keddad, MD, Study Director — PierreFabre Medicamment
Locations (17):
- Czechia (3):
  - Karlovy Vary
  - Prague
  - Praha 5 - Motol
- Budapest, Hungary
- Italy (5):
  - Augusta
  - Brescia
  - Foggia
  - Terni
  - Verona
- Poland (4):
  - Grodzisk Mazowiecki
  - Radom
  - Sandomierz
  - Warsaw
- Spain (4):
  - Barcelona
  - Madrid
  - Santiago de Compostela
  - Tarragona

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was planned to randomise a total of 152 patients. Due to low recruitment, the study recruitment was interrupted prematurely. Instead of 152 patients, 157 patients were screened and a total of 135 were finally randomised. 1 patient received no dose of the study treatment and was also not included in the analyses.
Pre-assignment Details: Patients were randomised after 1 to 4-week run-in period without study treatment.
Period: Overall Study
Arm/Group | F373280 | Placebo
Started | 67 | 67
Completed | 33 | 30
Not Completed | 34 | 37
Not completed — Adverse Event | 5 | 8
Not completed — Lack of Efficacy | 13 | 11
Not completed — Unsuccessful Electrical Cardioversion | 16 | 18

BASELINE CHARACTERISTICS:
Population: 134 patients were included in the Baseline Analysis Population (all randomised patients who received at least one dose of the study treatment).
Groups:
- F373280: 68 patients were randomised in the F373280 arm but one patient did not receive any dose of study treatment. 67 patients were also included in the analyses.
  1g of F373280: Oral administration, one capsule each evening with dinner.
- Placebo: 67 patients were randomised in the placebo arm. Placebo: Oral administration, one capsule each evening with dinner.
- Total: Total of all reporting groups
Arm/Group | F373280 | Placebo | Total
Number analyzed (Participants) | 67 | 67 | 134
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 33 | 62
  >=65 years | 38 | 34 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (9.7) | 65.9 (10.8) | 66.7 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 52 | 51 | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 67 | 67 | 134
Region of Enrollment [Number; unit: participants]
  Hungary | 13 | 13 | 26
  Czechia | 18 | 15 | 33
  Poland | 2 | 2 | 4
  Italy | 19 | 20 | 39
  Spain | 15 | 17 | 32
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (4.7) | 29.1 (4.9) | 28.8 (4.8)
Body surface area [Mean (Standard Deviation); unit: m^2] | 1.98 (0.19) | 2.02 (0.19) | 2.0 (0.19)

OUTCOME MEASURES:

1. Primary Outcome: Time to First Atrial Fibrillation (AF) Recurrence or Atrial Flutter Emergence Defined by the Time to First Episode of AF or Atrial Flutter Lasting for at Least 10 Minutes During the 20-week Follow-up After Visit 3 (Electrical Cardioversion (ECV) Visit).
Description: Time to first Atrial Fibrillation (AF) recurrence defined by the first episode of Atrial Fibrillation lasting for at least 10 minutes. AF recurrences or atrial flutter emergences: 7-day continuous electrocardiogram (ECG; 5-leads/2 or 3 channels) ambulatory recording (Holter ECG) between Visit 3 (Electrical Cardioversion Visit) and Visit 4 (Week 5). Then, the follow-up was documented using the Transtelephonic ECG monitor (TTEM): one transmission every two days from Week 9 to Week 24. For randomised patients with spontaneous cardioversion before Electrical Cardioversion, the recurrence of AF or the emergence of atrial flutter was assessed after Visit 3 (from Week 5). Moreover, during this TTEM period, if the patient experienced any AF or atrial flutter symptoms, it was recorded and documented using the TTEM.
Time Frame: from electrical cardioversion (Visit 3) to last follow-up visit (W24)
Population: The Full Analysis Set is composed of all randomised patients having received at least one dose of the study treatment and with a successful cardioversion observed at Visit 3; a successful cardioversion was defined as either spontaneous cardioversion before Visit 3 or successful Electrical Cardioversion performed at Visit 3.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | F373280 | Placebo
Number analyzed (Participants) | 52 | 49
days | 11.0 [6.0 to 45.0] | 16.0 [6.0 to 141.0]
Statistical Analysis 1: Comparison: F373280 vs Placebo; The primary criterion, time to first Atrial Fibrillation (AF) recurrence or atrial flutter emergence, was described using survival curves according to the Kaplan-Meier method, reporting the first and third quartiles (Q1, Q3), median, and 95% confidence interval. The time to first AF recurrence or atrial flutter emergence was compared between treatment groups using the Log rank test. Hazard ratios and 95% confidence intervals were estimated with the Cox regression model; Test type: Superiority; p = 0.5749, Log Rank; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.71 to 1.85]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the visit 2 to the last visit (Visit 9 Week 24).
Arm/Group | F373280 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/67 | 0/67
Serious Adverse Events (participants affected / at risk) | 5/67 | 1/67
Other Adverse Events (participants affected / at risk) | 41/67 | 38/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F373280 (N=67) | Placebo (N=67)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Cardiac disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F373280 (N=67) | Placebo (N=67)
Orthostatic hypotension (Vascular disorders) | 24 (33) | 20 (24)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypertension (Vascular disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 4 (4)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 5 (5)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Oedema peripheral (Cardiac disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1)
International normalised ratio decreased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-11-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT01831856/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT01831856/SAP_001.pdf